CLINICAL TRIAL: NCT01538446
Title: The ANTARCTIC Study - Assessment of a Normal Versus Tailored Dose of Prasugrel After Stenting in Patients Aged > 75 Years to Reduce the Composite of Bleeding, Stent Thrombosis and Ischemic Complications
Brief Title: Tailored Antiplatelet Therapy Versus Recommended Dose of Prasugrel
Acronym: ANTARCTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Eli Lilly and Company (Industry); Daiichi Sankyo (Industry); Allies in Cardiovascular Trials Initiatives and Organized (Other); Accumetrics, Inc. (Industry); Stentys (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110101
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Elderly; Acute coronary syndrome; Percutaneous coronary intervention; Prasugrel; Platelet function test
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Monitoring Arm (Experimental): Monitoring Arm: dose adjustment of prasugrel with down-adjustment of the dose of prasugrel in high responders and up-adjustment of the dose of prasugrel in low responders
  Interventions: Drug: Modification of Prasugrel based on a biological assay; Device: Verify Now
- 2: Conventional Arm (Active Comparator): Conventional Arm: fixed dose of prasugrel 5 mg
  Interventions: Drug: prasugrel / clopidogrel

INTERVENTIONS:
Drug: Modification of Prasugrel based on a biological assay — Monitoring with VerifyNow P2Y12, 2 weeks after initiation of 5 mg of maintenance dose of prasugrel, reduction of antiplatelet therapy if there is high on-treatment platelet inhibition (HPI) or increase in dosing if there is high on-treatment platelet reactivity (HPR) Device: VerifyNow point of care assay VerifyNow (ACCUMETRICS San Diego USA)
  Arms: 1: Monitoring Arm
Drug: prasugrel / clopidogrel — fixed dose of prasugrel 5 mg
  Arms: 2: Conventional Arm
Device: Verify Now — Monitoring with VerifyNow P2Y12, 2 weeks after initiation of 5 mg of maintenance dose of prasugrel, reduction of antiplatelet therapy if there is high on-treatment platelet inhibition (HPI) or increase in dosing if there is high on-treatment platelet reactivity (HPR) Device: VerifyNow point of care assay VerifyNow (ACCUMETRICS San Diego USA)
  Arms: 1: Monitoring Arm

SUMMARY:
The purpose of this study is to demonstrate the superiority of a strategy of platelet monitoring (Monitoring Arm) with down-adjustment of the dose of prasugrel in high responders and up-adjustment of the dose of prasugrel in low responders as compared to a more conventional strategy of a fixed dose of 5 mg to every patient without monitoring (Conventional Arm) as measured by a reduction in the composite endpoint of, cardiovascular (CV) death, myocardial infarction (MI) , stroke, stent thrombosis (ARC definition type "definite"), urgent revascularisation or bleeding (BARC definition type 2, 3 or 5).

DETAILED DESCRIPTION:
Objective: To demonstrate the superiority of a strategy of platelet monitoring (Monitoring Arm) with down-adjustment of the dose of prasugrel in high responders and up-adjustment of the dose of prasugrel in low responders as compared to a more conventional strategy of a fixed dose of 5 mg to every patient without monitoring (Conventional Arm).Rationale: Prasugrel 10 mg is superior to clopidogrel in patients with acute coronary syndrome treated by percutaneous coronary intervention, reducing significantly the rates of ischemic events. Elderly patients appear to be at higher risk of bleeding events and pharmacokinetic data suggests that elderly patients are exposed to a higher concentration of the active metabolite of prasugrel. A reduced dose of 5 mg of prasugrel is therefore proposed to these patients to limit the risk of bleeding. On the other hand, the elderly have also a higher ischemic risk and higher levels of platelet aggregation under treatment than younger patients and may deserve stronger protection from antiplatelet therapy. Platelet function testing appears to be of particular interest in patients at high risk of both ischemic and bleeding events like the elderly. Too intense platelet inhibition may expose the elderly patients to an excessive bleeding risk. Too low platelet inhibition may expose them to recurrent cardiovascular ischemic events. The possibility of bedside monitoring of oral antiplatelet therapy offers the opportunity of tailoring prasugrel therapy in elderly patients to optimize their risk/benefit ratio. Such strategy has never been evaluated in a randomized and adequately powered study. Population: Acute coronary syndrome (STEMI and NSTEMI) treated by PCI-stent (bare metal stent or drug eluting stent) in patients aged 75 ≥ year. Methods: Monitoring with VerifyNow P2Y12, 2 weeks after initiation of 5 mg of maintenance dose of prasugrel, reduction of antiplatelet therapy if there is high on-treatment platelet inhibition (HPI) or increase in dosing if there is high on-treatment platelet reactivity (HPR). Patients will be monitored again 2 weeks later, only if they do not meet the Verifynow P2Y12 targets at the first assessment. Primary endpoint net clinical benefit at 12 months:Composite of Cardiovascular death, myocardial infarction, stroke, urgent revascularisation, stent thrombosis and bleedings according to the BARC definitions (type 2, 3 or 5) Centers: Approximately 40 French high volume PCI centers

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome (STEMI and NSTEMI) treated by PCI
* Stent (bare metal stent or drug eluting stent) regardless of the regime of thienopyridines administered before randomisation
* Age ≥ 75 years.
* Aspirin dose of 75 mg will be recommended but study authorizes doses ranging from 75-160 mg
* Ability to understand and to comply with the study protocol.
* Written informed consent

Exclusion Criteria:

* Prior history of ischemic or hemorrhagic stroke or transient ischemic attack, or sub-arachnoids haemorrhage
* Have received fibrinolytic therapy within 48 hours of entry or randomisation into the study
* Are receiving vitamin K antagonist
* Concomitant medical illness (terminal malignancy) that is associated with reduced survival over the expected study treatment period.
* History of intolerance or allergy to ASA or approved thienopyridines (ticlopidine, clopidogrel, or prasugrel)
* Have active pathological bleeding or history of bleeding diathesis
* Thrombocytopenia < 100 000 µL
* Severe hepatic impairment (Child Pugh class C).
* Have a condition associated with poor treatment compliance, including dementia or mental illness

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 880 (Actual)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Composite of Cardiovascular death, myocardial infarction, stroke, urgent revascularisation, stent thrombosis and bleedings according to the BARC definitions (type 2, 3 or 5) through 12 months of randomisation | through 12 months of randomisation
  Composite of Cardiovascular death, myocardial infarction, stroke, urgent revascularisation, stent thrombosis and bleedings according to the BARC definitions (type 2, 3 or 5) through 12 months of randomisation

SECONDARY OUTCOMES:
Evaluation of the benefice of prasugrel adjustment on the composite ischemic endpoint of cardiovascular (CV) death, MI, definite stent thrombosis and Urgent revascularisation through 12 months of randomisation | through 12 months of randomisation
  The key secondary objective is to evaluate the benefice of prasugrel adjustment on the composite ischemic endpoint of cardiovascular (CV) death, MI, definite stent thrombosis and Urgent revascularisation through 12 months of randomisation
CV death, MI, stroke through 12 months of randomisation | through 12 months of randomisation
CV death, MI, stroke or Urgent Revascularization through 12 months of randomisation | through 12 months of randomisation
CV death: any death | 12 months after randomization
Any death or resuscitated cardiac death | 12 months after randomization
CV death or MI | 12 months after randomization
Definite stent thrombosis (ARC definition) | 12 months after randomization
All types of bleeding according to the BARC definitions 1, 2, 3, 4, 5 | 12 months after randomization
BARC Bleeding of type 2, 3 or 5 | 12 months after randomization
Bleeding TIMI major through 12 months of randomisation | through 12 months of randomisation
GUSTO severe or moderate bleeding | 12 months after randomization
STEEPLE bleeding definitions (major, minor or both) | 12 months after randomization
ISTH bleeding definitions (major and clinically relevant non major) | 12 months after randomization
Bleeding TIMI minor | 12 months after randomization
Bleeding TIMI minimal | 12 months after randomization
Bleeding TIMI major, minor and combination | 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MONTALESCOT, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - CHU Caremeau à Nimes - Service de Cardiologie, Nîmes
  - ACTION study group - Institut de Cardiologie- Hôpital la Pitié Salpêtrière, Paris

REFERENCES:
- [Result] Cayla G, Cuisset T, Silvain J, Leclercq F, Manzo-Silberman S, Saint-Etienne C, Delarche N, Bellemain-Appaix A, Range G, El Mahmoud R, Carrie D, Belle L, Souteyrand G, Aubry P, Sabouret P, du Fretay XH, Beygui F, Bonnet JL, Lattuca B, Pouillot C, Varenne O, Boueri Z, Van Belle E, Henry P, Motreff P, Elhadad S, Salem JE, Abtan J, Rousseau H, Collet JP, Vicaut E, Montalescot G; ANTARCTIC investigators. Platelet function monitoring to adjust antiplatelet therapy in elderly patients stented for an acute coronary syndrome (ANTARCTIC): an open-label, blinded-endpoint, randomised controlled superiority trial. Lancet. 2016 Oct 22;388(10055):2015-2022. doi: 10.1016/S0140-6736(16)31323-X. Epub 2016 Aug 28. PMID 27581531
- [Derived] Lattuca B, Cayla G, Silvain J, Cuisset T, Leclercq F, Manzo-Silberman S, Saint-Etienne C, Delarche N, El Mahmoud R, Carrie D, Souteyrand G, Kerneis M, Hauguel-Moreau M, Zeitouni M, Guedeney P, Diallo A, Collet JP, Vicaut E, Montalescot G; ACTION Study Group. Bleeding in the Elderly: Risk Factors and Impact on Clinical Outcomes After an Acute Coronary Syndrome, a Sub-study of the Randomized ANTARCTIC Trial. Am J Cardiovasc Drugs. 2021 Nov;21(6):681-691. doi: 10.1007/s40256-021-00468-8. Epub 2021 Jun 30. PMID 34191259
- [Derived] Cayla G, Cuisset T, Silvain J, Henry P, Leclercq F, Carrie D, Etienne CS, Belle L, Range G, Pouillot C, Varenne O, Van Belle E, Boueri Z, Motreff P, Elhadad S, Delarche N, El Mahmoud R, Vicaut E, Collet JP, Montalescot G; ANTARCTIC investigators. Platelet function monitoring in elderly patients on prasugrel after stenting for an acute coronary syndrome: design of the randomized antarctic study. Am Heart J. 2014 Nov;168(5):674-81. doi: 10.1016/j.ahj.2014.07.026. Epub 2014 Aug 7. PMID 25440795